CLINICAL TRIAL: NCT00739297
Title: A Phase Ib Randomized, Placebo-Controlled Clinical Trial to Study the Safety and Bronchodilatory Effect of MK0476 in Patients With Chronic Asthma
Brief Title: The Safety and Effectiveness of MK0476 (Montelukast) in Patients With Chronic Asthma (0476-388)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-388; MK0476-388; 2008_542
Record Dates: First submitted 2008-08-19; First posted 2008-08-21 (Estimated); Results first posted 2010-04-09 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2022-02

CONDITIONS: Chronic Asthma
Keywords: Chronic asthma
MeSH Terms: interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Placebo Comparator): montelukast Placebo
  Interventions: Drug: Comparator: montelukast; Drug: Comparator: placebo
- 2 (Experimental): montelukast
  Interventions: Drug: Comparator: montelukast
- 3 (Experimental): montelukast
  Interventions: Drug: Comparator: montelukast
- 4 (Experimental): montelukast
  Interventions: Drug: Comparator: montelukast

INTERVENTIONS:
Drug: Comparator: montelukast — 5 Period, Cross-over, Dose-Ranging study. Period I: no treatment. Periods II-V: Single-dose administration of inhaled montelukast (using doses as low as 25 mcg, to as high as 1000 mcg), or montelukast placebo. Two puffs of albuterol or albuterol placebo will be given four hours after montelukast/montelukast placebo.
  Other Names: SINGULAIR®, PROAIR® HFA
Drug: Comparator: placebo — 5 Period, Cross-over, Dose-Ranging study. Period I: no treatment. Periods II-V: Single-dose administration of inhaled montelukast (using doses as low as 25 mcg, to as high as 1000 mcg), or montelukast placebo. Two puffs of albuterol or albuterol placebo will be given four hours after montelukast/montelukast placebo.
  Arms: 1

SUMMARY:
This study will test the safety and effectiveness of a range of doses of MK0476 (montelukast) compared to placebo on improved lung function in patients with chronic asthma.

ELIGIBILITY:
Inclusion Criteria:

* A person is 15 to 65 years of age. A person has had chronic asthma for at least one year

Exclusion Criteria:

* A person is a smoker or has smoked more that a pack a day for more than 10 years before stopping
* A person has other lung disorders such as COPD (chronic obstructive pulmonary disorder)

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2008-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Philip G, Pedinoff A, Vandormael K, Tymofyeyev Y, Smugar SS, Reiss TF, Korenblat PE. A phase I randomized, placebo-controlled, dose-exploration study of single-dose inhaled montelukast in patients with chronic asthma. J Asthma. 2010 Dec;47(10):1078-84. doi: 10.3109/02770903.2010.520100. Epub 2010 Nov 3. PMID 20936994

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 6 centers in the United States between July and December 2008.
Pre-assignment Details: 117 participants were screened; 49 were excluded. Randomized patients met the following criteria during the prestudy period: FEV1 (Forced expiratory volume in one second) 50-85% predicted while withholding short-acting beta agonist (SABA) and reversibility of airway obstruction >12% following SABA at Visits 1 and 2.
Groups:
- Placebo: Patients are randomized to receive placebo for montelukast on either Intervention I (Visit 3), Intervention II (Visit 5), Intervention III (Visit 7) or Intervention IV (Visit 9). At all interventions, either albuterol or placebo for albuterol is administered 4 hours after placebo for montelukast. During the washout periods separating the intervention periods, patients received no study treatment (i.e., patients did not receive montelukast or placebo treatment).
- 25 mcg Montelukast: Patients are randomized to receive montelukast 25 mcg (microgram) on either Intervention I (Visit 3), Intervention II (Visit 5), Intervention III (Visit 7) or Intervention IV (Visit 9). At all interventions either albuterol or placebo for albuterol is administered 4 hours after montelukast 25 mcg. During the washout periods separating the intervention periods, patients received no study treatment (i.e., patients did not receive montelukast or placebo treatment).
- 100 mcg Montelukast: Patients are randomized to receive montelukast 100 mcg on either Intervention I (Visit 3), Intervention II (Visit 5), Intervention III (Visit 7) or Intervention IV (Visit 9). At all interventions either albuterol or placebo for albuterol is administered 4 hours after montelukast 100 mcg. During the washout periods separating the intervention periods, patients received no study treatment (i.e., patients did not receive montelukast or placebo treatment).
- 250 mcg Montelukast: Patients are randomized to receive montelukast 250 mcg on either Intervention I (Visit 3), Intervention II (Visit 5), Intervention III (Visit 7) or Intervention IV (Visit 9). At all interventions either albuterol or placebo for albuterol is administered 4 hours after montelukast 250 mcg. During the washout periods separating the intervention periods, patients received no study treatment (i.e., patients did not receive montelukast or placebo treatment).
- 500 mcg Montelukast: Patients are randomized to receive montelukast 500 mcg on either Intervention I (Visit 3), Intervention II (Visit 5), Intervention III (Visit 7) or Intervention IV (Visit 9). At all interventions either albuterol or placebo for albuterol is administered 4 hours after montelukast 500 mcg. During the washout periods separating the intervention periods, patients received no study treatment (i.e., patients did not receive montelukast or placebo treatment).
- 1000 mcg Montelukast: Patients are randomized to receive montelukast 1000 mcg on either Intervention I (Visit 3), Intervention II (Visit 5), Intervention III (Visit 7) or Intervention IV (Visit 9). At all interventions either albuterol or placebo for albuterol is administered 4 hours after montelukast 1000 mcg. During the washout periods separating the intervention periods, patients received no study treatment (i.e., patients did not receive montelukast or placebo treatment).
- Total: Consistent with the "incomplete-block" design of this study, 6 treatments (placebo and 5 active-dose levels) were administered during only 4 treatment periods. In other words, in this 4-period crossover design, no patient received all 6 treatments and thus some treatments were not
  received by all of the patients. Therefore, the TOTAL number of participants across ALL the dose levels provides the best metric to follow the consistency of patient flow from one treatment period to the next treatment period.
Period: First Intervention (Visit 3 to Visit 4)
Arm/Group | Placebo | 25 mcg Montelukast | 100 mcg Montelukast | 250 mcg Montelukast | 500 mcg Montelukast | 1000 mcg Montelukast | Total
Started | 17 | 11 | 6 | 19 | 6 | 9 | 68
Completed | 17 | 11 | 6 | 19 | 6 | 9 | 68
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: First Washout Period of 4-7 Days
Arm/Group | Placebo | 25 mcg Montelukast | 100 mcg Montelukast | 250 mcg Montelukast | 500 mcg Montelukast | 1000 mcg Montelukast | Total
Started | 17 | 11 | 6 | 19 | 6 | 9 | 68
Completed | 17 | 11 | 6 | 17 | 6 | 9 | 66
Not Completed | 0 | 0 | 0 | 2 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0 | 0 | 2
Period: Second Intervention (Visit 5 to Visit 6)
Arm/Group | Placebo | 25 mcg Montelukast | 100 mcg Montelukast | 250 mcg Montelukast | 500 mcg Montelukast | 1000 mcg Montelukast | Total
Started | 18 | 8 | 10 | 14 | 6 | 10 | 66
Completed | 18 | 8 | 10 | 14 | 6 | 10 | 66
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Washout Period of 4-7 Days
Arm/Group | Placebo | 25 mcg Montelukast | 100 mcg Montelukast | 250 mcg Montelukast | 500 mcg Montelukast | 1000 mcg Montelukast | Total
Started | 18 | 8 | 10 | 14 | 6 | 10 | 66
Completed | 18 | 8 | 10 | 14 | 6 | 10 | 66
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (Visit 7 to Visit 8)
Arm/Group | Placebo | 25 mcg Montelukast | 100 mcg Montelukast | 250 mcg Montelukast | 500 mcg Montelukast | 1000 mcg Montelukast | Total
Started | 16 | 12 | 6 | 18 | 6 | 8 | 66
Completed | 16 | 12 | 6 | 18 | 6 | 8 | 66
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Washout Period of 4-7 Days
Arm/Group | Placebo | 25 mcg Montelukast | 100 mcg Montelukast | 250 mcg Montelukast | 500 mcg Montelukast | 1000 mcg Montelukast | Total
Started | 16 | 12 | 6 | 18 | 6 | 8 | 66
Completed | 16 | 12 | 6 | 18 | 6 | 8 | 66
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Fourth Intervention(Visit 9 to Visit 10)
Arm/Group | Placebo | 25 mcg Montelukast | 100 mcg Montelukast | 250 mcg Montelukast | 500 mcg Montelukast | 1000 mcg Montelukast | Total
Started | 16 | 11 | 8 | 15 | 7 | 9 | 66
Completed | 16 | 11 | 8 | 15 | 7 | 8 | 65
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Patient unable to attend last visit | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Combined participants from all arms.
Arm/Group | All Participants
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 36
FEV1 (Forced Expiratory Volume in One Second) [Mean (Standard Deviation); unit: L (Liter)] | 2.44 (0.63)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in FEV1 Over 4 Hours
Description: FEV1 measurements taken at 0 (=baseline), 10, 20, 30, 45, 60, 120, 180 and 240 minutes contributed to the average change from baseline over 4 hours. The number of minutes between consecutive measurements was used as weighting factor. The time-weighted average change was standardized by dividing by the time associated with the last measurement.
Time Frame: 0 (=baseline) to 4 hours after treatment with montelukast
Population: Full analysis set (FAS) population which included all randomized patients who took at least one dose of post randomization study drug (Montelukast or placebo) at either of the intervention visits and had a measurement for analysis available in at least one treatment period of the cross-over design.
Measure: Least Squares Mean (95% Confidence Interval); unit: L (Liter)
Arm/Group | Placebo | 25 mcg Montelukast | 100 mcg Montelukast | 250 mcg Montelukast | 500 mcg Montelukast | 1000 mcg Montelukast
Number analyzed (Participants) | 67 | 42 | 30 | 66 | 25 | 36
L (Liter) | 0.03 [-0.03 to 0.10] | 0.07 [0.00 to 0.14] | 0.13 [0.06 to 0.20] | 0.10 [0.04 to 0.16] | 0.09 [0.01 to 0.16] | 0.12 [0.05 to 0.19]
Statistical Analysis 1: Comparison: Placebo vs 25 mcg Montelukast; Test type: Superiority or Other; Difference in Least-Squares Means = 0.04, 95% CI [-0.01 to 0.08] — Mixed effects model with terms for treatment (including dose of montelukast), period and baseline covariate
Statistical Analysis 2: Comparison: Placebo vs 100 mcg Montelukast; Test type: Superiority or Other; Difference in Least-Squares Means = 0.10, 95% CI [0.04 to 0.15] — Mixed effects model with terms for treatment (including dose of montelukast), period and baseline covariate
Statistical Analysis 3: Comparison: Placebo vs 250 mcg Montelukast; Test type: Superiority or Other; Difference in Least-Squares Means = 0.06, 95% CI [0.02 to 0.11] — Mixed effects model with terms for treatment (including dose of montelukast), period and baseline covariate
Statistical Analysis 4: Comparison: Placebo vs 500 mcg Montelukast; Test type: Superiority or Other; Difference in Least-Squares Means = 0.05, 95% CI [-0.01 to 0.11] — Mixed effects model with terms for treatment (including dose of montelukast), period and baseline covariate
Statistical Analysis 5: Comparison: Placebo vs 1000 mcg Montelukast; Test type: Superiority or Other; Difference in Least-Squares Means = 0.08, 95% CI [0.04 to 0.13] — Mixed effects model with terms for treatment (including dose of montelukast), period and baseline covariate

2. Secondary Outcome: Change From Baseline in FEV1 Over 90 Minutes After Albuterol/Placebo Administration
Description: FEV1 measurements taken at 0 (=baseline), 15, 30, 60, and 90 minutes after albuterol/placebo administration contributed to the average change from baseline over 90 minutes. The number of minutes between consecutive measurements was used as weighting factor. The time-weighted average change was standardized by dividing by the time associated with the last measurement.
Time Frame: 4 hours (equals time point at which albuterol or albuterol placebo is administered) to 5.5 hours after treatment with montelukast
Population: Full analysis set (FAS) population which included all randomized patients who took at least one dose of post randomization study drug (albuterol or matching placebo) 4 hours after treatment with montelukast at either of the intervention visits and had a measurement for analysis available in at least one treatment period of the cross-over design.
Measure: Least Squares Mean (95% Confidence Interval); unit: L
Groups:
- Montelukast+Albuterol: Montelukast (data for each patient are pooled across all 3 of the active doses received by that patient) +Albuterol (data for each patient are pooled across all 3 administrations of active albuterol, as added to active montelukast)
- Montelukast+ Placebo: Montelukast (data for each patient are pooled across all 3 of the active doses received by that patient) +Placebo for Albuterol (data for each patient are pooled across all 3 administrations of placebo for albuterol, as added to active montelukast)
Arm/Group | Montelukast+Albuterol | Montelukast+ Placebo
Number analyzed (Participants) | 26 | 41
L | 0.34 [0.22 to 0.45] | 0.15 [0.06 to 0.24]
Statistical Analysis 1: Comparison: Montelukast+Albuterol vs Montelukast+ Placebo; Test type: Superiority or Other; Difference in Least-Squares Means = 0.19, 95% CI [0.04 to 0.34] — Repeated measures model with terms for treatment (Albuterol/Placebo), dose, treatment-by-dose interaction and baseline FEV1

3. Other Pre Specified Outcome: Change From Baseline in FEV1 at 8 Hours After Treatment With Montelukast
Description: Average change from baseline in FEV1 at 8 hours after single dose montelukast administration.
Time Frame: 0 (baseline) and 8 hours after treatment with montelukast
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: L
Arm/Group | Placebo | 25 mcg Montelukast | 100 mcg Montelukast | 250 mcg Montelukast | 500 mcg Montelukast | 1000 mcg Montelukast
Number analyzed (Participants) | 67 | 42 | 30 | 66 | 24 | 35
L | 0.06 [-0.02 to 0.14] | 0.11 [0.03 to 0.20] | 0.13 [0.04 to 0.23] | 0.11 [0.03 to 0.19] | 0.12 [0.02 to 0.22] | 0.14 [0.05 to 0.23]
Statistical Analysis 1: Comparison: Placebo vs 25 mcg Montelukast; Test type: Superiority or Other; Difference in Least-Squares Means = 0.06, 95% CI [-0.01 to 0.12] — Mixed effects model with terms for treatment (including dose of montelukast), period and baseline covariate
Statistical Analysis 2: Comparison: Placebo vs 100 mcg Montelukast; Test type: Superiority or Other; Difference in Least-Squares Means = 0.07, 95% CI [-0.00 to 0.15] — Mixed effects model with terms for treatment (including dose of montelukast), period and baseline covariate
Statistical Analysis 3: Comparison: Placebo vs 250 mcg Montelukast; Test type: Superiority or Other; Difference in Least-Squares Means = 0.05, 95% CI [-0.01 to 0.11] — Mixed effects model with terms for treatment (including dose of montelukast), period and baseline covariate
Statistical Analysis 4: Comparison: Placebo vs 500 mcg Montelukast; Test type: Superiority or Other; Difference in Least-Squares Means = 0.06, 95% CI [-0.03 to 0.14] — Mixed effects model with terms for treatment (including dose of montelukast), period and baseline covariate
Statistical Analysis 5: Comparison: Placebo vs 1000 mcg Montelukast; Test type: Superiority or Other; Difference in Least-Squares Means = 0.08, 95% CI [0.01 to 0.15] — Mixed effects model with terms for treatment (including dose of montelukast), period and baseline covariate

4. Other Pre Specified Outcome: Change From Baseline in FEV1 at 24 Hours After Treatment With Montelukast
Description: Average change from baseline in FEV1 at 24 hours after single dose montelukast administration.
Time Frame: 0 (baseline) and 24 hours after treatment with montelukast
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: L
Arm/Group | Placebo | 25 mcg Montelukast | 100 mcg Montelukast | 250 mcg Montelukast | 500 mcg Montelukast | 1000 mcg Montelukast
Number analyzed (Participants) | 67 | 42 | 29 | 66 | 25 | 36
L | 0.02 [-0.06 to 0.09] | 0.05 [-0.03 to 0.13] | 0.10 [0.01 to 0.19] | 0.06 [-0.01 to 0.13] | 0.08 [-0.01 to 0.18] | 0.09 [0.01 to 0.18]
Statistical Analysis 1: Comparison: Placebo vs 25 mcg Montelukast; Test type: Superiority or Other; Difference in Least-Squares Means = 0.04, 95% CI [-0.03 to 0.10] — Mixed effects model with terms for treatment (including dose of montelukast), period and baseline covariate
Statistical Analysis 2: Comparison: Placebo vs 100 mcg Montelukast; Test type: Superiority or Other; Difference in Least-Squares Means = 0.09, 95% CI [0.01 to 0.17] — Mixed effects model with terms for treatment (including dose of montelukast), period and baseline covariate
Statistical Analysis 3: Comparison: Placebo vs 250 mcg Montelukast; Test type: Superiority or Other; Difference in Least-Squares Means = 0.05, 95% CI [-0.01 to 0.10] — Mixed effects model with terms for treatment (including dose of montelukast), period and baseline covariate
Statistical Analysis 4: Comparison: Placebo vs 500 mcg Montelukast; Test type: Superiority or Other; Difference in Least-Squares Means = 0.07, 95% CI [-0.02 to 0.15] — Mixed effects model with terms for treatment (including dose of montelukast), period and baseline covariate
Statistical Analysis 5: Comparison: Placebo vs 1000 mcg Montelukast; Test type: Superiority or Other; Difference in Least-Squares Means = 0.08, 95% CI [0.01 to 0.15] — Mixed effects model with terms for treatment (including dose of montelukast), period and baseline covariate

ADVERSE EVENTS:
Arm/Group | Placebo | 25 mcg Montelukast | 100 mcg Montelukast | 250 mcg Montelukast | 500 mcg Montelukast | 1000 mcg Montelukast
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/41 | 0/30 | 0/66 | 0/25 | 0/36
Other Adverse Events (participants affected / at risk) | 4/67 | 1/41 | 0/30 | 3/66 | 3/25 | 0/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=67) | 25 mcg Montelukast (N=41) | 100 mcg Montelukast (N=30) | 250 mcg Montelukast (N=66) | 500 mcg Montelukast (N=25) | 1000 mcg Montelukast (N=36)
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.